CLINICAL TRIAL: NCT00338650
Title: A Multi-Center, Open-Label Treatment Protocol of the Human Anti-TNF Monoclonal Antibody Adalimumab in Patients With Moderate to Severe Crohn's Disease With Previous Exposure to Infliximab
Brief Title: Treatment of the Human Anti-TNF Monoclonal Antibody Adalimumab in Moderate to Severe Crohn's Disease With Previous Exposure to Infliximab (CHOICE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M06-808; CHOICE
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

INTERVENTIONS:
Drug: adalimumab

SUMMARY:
The primary objective of this study is to make adalimumab available to patients suffering from moderately to severely active Crohn's Disease who have failed to respond to, lost response to, or are intolerant to infliximab, and to evaluate safety

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with moderate to severe Crohn's Disease.
* Failed prior infliximab therapy.
* Patient is judged to be in generally good health as determined by the principal investigator.

Exclusion Criteria:

* Previous treatment with adalimumab.
* Patient considered by the investigator, for any reason, to be an unsuitable candidate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2006-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
AEs, laboratory data, physical examinations and vital signs

SECONDARY OUTCOMES:
Efficacy variables will be assessed from Outcomes Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Paperiello, Study Director — Abbott
Locations (77):
- United States (77):
  - Birmingham, Alabama
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Roseville, California
  - San Francisco, California
  - Englewood, Colorado
  - Wheat Ridge, Colorado
  - Bridgeport, Connecticut
  - Hamden, Connecticut
  - Clearwater, Florida
  - Gainesville, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Conyers, Georgia
  - Marietta, Georgia
  - Savannah, Georgia
  - Arlington Heights, Illinois
  - Moline, Illinois
  - Rockford, Illinois
  - Columbus, Indiana
  - Indianapolis, Indiana
  - Clive, Iowa
  - Davenport, Iowa
  - Overland Park, Kansas
  - Topeka, Kansas
  - Lexington, Kentucky
  - Annapolis, Maryland
  - Chevy Chase, Maryland
  - Lutherville, Maryland
  - Silver Spring, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Troy, Michigan
  - Plymouth, Minnesota
  - Picayune, Mississippi
  - Kansas City, Missouri
  - Mexico, Missouri
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Egg Harbor, New Jersey
  - Glen Ridge, New Jersey
  - Manalapan, New Jersey
  - Great Neck, New York
  - Lake Success, New York
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Jacksonville, North Carolina
  - Rocky Mount, North Carolina
  - Wilmington, North Carolina
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Warren, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Beaver Falls, Pennsylvania
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sayre, Pennsylvania
  - Columbia, South Carolina
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Austin, Texas
  - South Ogden, Utah
  - Norfolk, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Vancouver, Washington
  - Milwaukee, Wisconsin
  - Monroe, Wisconsin

REFERENCES:
- [Derived] Lichtiger S, Binion DG, Wolf DC, Present DH, Bensimon AG, Wu E, Yu AP, Cardoso AT, Chao J, Mulani PM, Lomax KG, Kent JD. The CHOICE trial: adalimumab demonstrates safety, fistula healing, improved quality of life and increased work productivity in patients with Crohn's disease who failed prior infliximab therapy. Aliment Pharmacol Ther. 2010 Nov;32(10):1228-39. doi: 10.1111/j.1365-2036.2010.04466.x. Epub 2010 Sep 28. PMID 20955442